CLINICAL TRIAL: NCT00463437
Title: Booster Vaccination With Pneumococcal Vaccine GSK1024850A, a DTPa-Combined and MenC or Hib-MenC Vaccines
Brief Title: Pneumococcal Vaccine Booster Study in Healthy Children 11-18 Months Old Previously Primed With the Same Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109507; 2006-005733-38 (EudraCT Number)
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B; Acellular Pertussis; Tetanus; Poliomyelitis; Diphtheria; Streptococcus Pneumoniae Vaccines
Keywords: Fever.; Meningococcal disease.; Pneumococcal disease.; Meningococcal vaccine.; Pneumococcal vaccine.; Immunogenicity.; Booster vaccination.; Safety.
MeSH Terms: conditions — Hepatitis B; Tetanus; Poliomyelitis; Diphtheria; Fever; Meningococcal Infections; Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; serogroup C meningococcal conjugate vaccine

ARMS (4):
- GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ (Experimental): Subjects receiving a booster dose of pneumococcal conjugate vaccine GSK1024850A co-administered with GSK Biologicals' DTPa-combined vaccine (Infanrix™ hexa in Germany & Poland and Infanrix™ IPV Hib in Spain) and Wyeth's Men-C conjugate vaccine (Meningitec™) at 11-18 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Infanrix hexa; Biological: Infanrix IPV Hib; Biological: Meningitec
- GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ (Experimental): Subjects receiving a booster dose of pneumococcal conjugate vaccine GSK1024850A co-administered with GSK Biologicals' DTPa-combined vaccine (Infanrix™ hexa in Germany & Poland and Infanrix™ IPV Hib in Spain) and Baxter's Men-C conjugate vaccine (NeisVac-C™) at 11-18 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Infanrix hexa; Biological: Infanrix IPV Hib; Biological: NeisVac-C
- GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ (Experimental): Subjects receiving a booster dose of pneumococcal conjugate vaccine GSK1024850A co-administered with DTPa-combined vaccine (Infanrix™ penta in Germany & Poland and Infanrix™ IPV in Spain) and GSK Biologicals' combined Hib-MenC vaccine (Menitorix™) at 11-18 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Infanrix penta; Biological: Infanrix IPV; Biological: Menitorix
- Prevenar™ + Menitorix™ (Active Comparator): Subjects receiving a booster dose of Wyeth's pneumococcal conjugate vaccine (Prevenar™) co-administered with DTPa-combined vaccine (Infanrix™ penta in Germany & Poland and Infanrix™ IPV in Spain) and GSK Biologicals' combined Hib-MenC vaccine (Menitorix™) at 11-18 months of age.
  Interventions: Biological: Prevenar; Biological: Infanrix penta; Biological: Infanrix IPV; Biological: Menitorix

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection, 1 dose.
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™; GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™; GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™
Biological: Prevenar — Intramuscular injection, 1 dose.
  Other Names: Pneumococcal conjugate vaccine (Wyeth Lederle).
  Arms: Prevenar™ + Menitorix™
Biological: Infanrix hexa — Intramuscular injection, 1 dose. In Germany and Poland.
  Other Names: DTPa-HBV-IPV/Hib (GSK Biologicals).
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™; GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™
Biological: Infanrix IPV Hib — Intramuscular injection, 1 dose. In Spain.
  Other Names: DTPa-IPV/Hib (GSK Biologicals).
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™; GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™
Biological: Infanrix penta — Intramuscular injection, 1 dose. In Germany and Poland.
  Other Names: DTPa-HBV-IPV (GSK Biologicals).
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™; Prevenar™ + Menitorix™
Biological: Infanrix IPV — Intramuscular injection, 1 dose. In Spain.
  Other Names: DTPa-IPV (GSK Biologicals)
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™; Prevenar™ + Menitorix™
Biological: Meningitec — Intramuscular injection, 1 dose.
  Other Names: Meningococcal C conjugate vaccine (Wyeth).
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™
Biological: NeisVac-C — Intramuscular injection, 1 dose.
  Other Names: Meningococcal C conjugate vaccine (Baxter).
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™
Biological: Menitorix — Intramuscular injection, 1 dose.
  Other Names: Combined Hib-MenC vaccine (GSK Biologicals).
  Arms: GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™; Prevenar™ + Menitorix™

SUMMARY:
The purpose of this study is to assess the safety in terms of fever (rectal temperature) higher than 39 degree Celcius (°C) and the immunogenicity in terms of antibody response following a booster vaccination with pneumococcal vaccine GSK1024850A at 11 to 18 months of age in children previously primed with the same vaccines including a pneumococcal conjugate vaccine co-administered with a diphtheria, tetanus, acellular pertussis (DTPa)-combined and meningococcal serogroup C (MenC) or combined meningococcal serogroup C and Haemophilus influenzae type b (Hib-MenC) vaccine.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00334334).

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 11-18 months of age at the time of the booster vaccination.
* A male or female who previously participated in study 107005 and received three doses of pneumococcal conjugate vaccine.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period (active phase and extended safety follow-up), in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within one month preceding the booster dose of study vaccines, or planned use during the entire study period
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the booster dose of study vaccines.
* Planned administration/administration of a vaccine not foreseen by the study protocol, during the period starting one month before the booster dose of study vaccines and up to the follow-up visit (one month after the booster dose of study vaccines).
* Administration of any pneumococcal, diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, MenC and/or Hib-MenC vaccines other than the study vaccines from study 107005.
* History of, or intercurrent, diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, meningococcal serogroup C disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or progressive neurological disease.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products within three months preceding the booster dose of study vaccines or planned administration during the active phase of the study (starting with the administration of the booster dose of study vaccines up to the follow-up visit one month after).

Ages: 11 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1437 (Actual)
Dates: Start 2007-04-25 (Actual); Primary Completion 2008-01-21 (Actual); Study Completion 2008-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- Germany (35):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bönnigheim, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Roding, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Niedernhausen, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Bodenheim, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gerolstein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Singwitz, Saxony
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin
- Poland (7):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Wola
- Spain (12):
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Montgat/Barcelona
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Sant Vicenç Dels Horts /Barcelona
  - GSK Investigational Site, Tona/Barcelona
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vélez-Málaga / Málaga

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=134

REFERENCES:
- [Background] Chevallier B, Vesikari T, Brzostek J, Knuf M, Bermal N, Aristegui J, Borys D, Cleerbout J, Lommel P, Schuerman L. Safety and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with routine childhood vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S109-18. doi: 10.1097/INF.0b013e318199f62d. PMID 19325447
- [Background] Knuf M, Szenborn L, Moro M, Petit C, Bermal N, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of routinely used childhood vaccines when coadministered with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S97-S108. doi: 10.1097/INF.0b013e318199f61b. PMID 19325452
- [Background] Wysocki J, Tejedor JC, Grunert D, Konior R, Garcia-Sicilia J, Knuf M, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with different neisseria meningitidis serogroup C conjugate vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S77-88. doi: 10.1097/INF.0b013e318199f609. PMID 19325450
- [Background] Silfverdal SA, Coremans V, Francois N, Borys D, Cleerbout J. Safety profile of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Expert Rev Vaccines. 2017 Feb;16(2):109-121. doi: 10.1586/14760584.2016.1164044. Epub 2016 Sep 30. PMID 26954689
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Started | 359 | 363 | 358 | 357
Completed | 355 | 352 | 352 | 350
Not Completed | 4 | 11 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™ | Total
Number analyzed (Participants) | 359 | 363 | 358 | 357 | 1437
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.3 (1.81) | 14.3 (1.74) | 14.3 (1.78) | 14.3 (1.78) | 14.3 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 176 | 195 | 171 | 724
  Male | 177 | 187 | 163 | 186 | 713

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Fever Above 39.0 Degree Celsius (°C)
Description: Fever was measured as rectal temperature.
Time Frame: During the 4-day (Day 0-3) period after the booster vaccination
Population: Analysis was performed on the Total vaccinated cohort from Pn-HibC and Pr-HibC Groups on subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 0 | 0 | 355 | 355
subjects |  |  | 11 | 8

2. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 4-day (Day 0-3) period after the booster vaccination
Population: Subjects from the Total Vaccinated cohort for whom data were available.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 356 | 357 | 355 | 355
subjects
  Pain | 196 | 195 | 193 | 165
  Redness | 194 | 183 | 186 | 173
  Swelling | 162 | 148 | 150 | 134

3. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever, irritability, and loss of appetite.
Time Frame: During the 4-day (Day 0-3) period after the booster vaccination
Population: Subjects from the Total Vaccinated cohort for whom data were available.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 356 | 357 | 355 | 355
subjects
  Drowsiness | 124 | 142 | 139 | 105
  Fever (≥ 38.0 °C) | 109 | 122 | 105 | 108
  Irritability | 170 | 190 | 191 | 157
  Loss of appetite | 101 | 99 | 112 | 93

4. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day (Day 0-30) period after the booster vaccination
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 359 | 363 | 358 | 357
subjects | 59 | 74 | 59 | 76

5. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 31-day (Day 0-30) period after the booster vaccination
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 359 | 363 | 358 | 357
subjects | 3 | 5 | 3 | 2

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: as for outcome 5
Time Frame: From the beginning of the study up to the end of the extended 6-month safety follow-up period
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 359 | 363 | 358 | 357
subjects | 15 | 9 | 13 | 13

7. Secondary Outcome: Number of Subjects With Vaccine Pneumococcal Serotype Antibody Concentrations Above the Cut-off Value
Description: Anti-pneumococcal antibody concentration cut-off value assessed was 0.05 microgram per milliliter (µg/mL).
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 158 | 158 | 160 | 153
subjects
  Anti-1 pre (n=150,152,149, 151) | 146 | 146 | 140 | 21
  Anti-1 post (n=158,152,160,151) | 158 | 152 | 160 | 28
  Anti-4 pre (n=153,156,150,153) | 152 | 156 | 147 | 150
  Anti-4 post (n=158,153,160,152) | 158 | 153 | 160 | 152
  Anti-5 pre (n=149,146,146,148) | 149 | 146 | 144 | 37
  Anti-5 post (n=157,153,160,150) | 157 | 153 | 160 | 64
  Anti-6B pre (n=151,155,150,151) | 149 | 153 | 144 | 137
  Anti-6B post (n=158,153,160,153) | 157 | 151 | 158 | 153
  Anti-7F pre (n=149,153,148,151) | 149 | 153 | 147 | 18
  Anti-7F post (n=158,152,160,151) | 158 | 152 | 160 | 25
  Anti-9V pre (n=149,155,149,152) | 149 | 154 | 149 | 152
  Anti-9V post (n=158,153,160,153) | 158 | 152 | 160 | 153
  Anti-14 pre (n=153,158,152,153) | 151 | 157 | 152 | 151
  Anti-14 post (n=158,153,160,153) | 158 | 153 | 160 | 153
  Anti-18C pre (n=151,153,145,151) | 149 | 151 | 145 | 151
  Anti-18C post (n=157,152,160,152) | 157 | 152 | 160 | 152
  Anti-19F pre (n=143,146,139,150) | 143 | 146 | 139 | 143
  Anti-19F post (n=158,151,160,152) | 158 | 151 | 160 | 152
  Anti-23F pre (n=152,156,150,153) | 149 | 153 | 144 | 141
  Anti-23F post (n=158,153,160,153) | 158 | 152 | 158 | 153

8. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes Above the Cut-off Value
Description: Cut-off value for opsonophagocytic activity against pneumococcal antibody assessed was ≥ 8.
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, 23F.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 145 | 145 | 146 | 143
subjects
  Opsono-1 pre (n=144,145,141,143) | 46 | 39 | 41 | 8
  Opsono-1 post (n=140,139,140,137) | 132 | 133 | 127 | 12
  Opsono-4 pre (n=104,121,112,109) | 61 | 67 | 61 | 73
  Opsono-4 post (n=137,134,140,135) | 137 | 134 | 140 | 135
  Opsono-5 pre (n=116,114,117,124) | 77 | 71 | 72 | 3
  Opsono-5 post (n=124,130,136,127) | 121 | 127 | 131 | 4
  Opsono-6B pre (n=133,132,133,137) | 75 | 60 | 75 | 67
  Opsono-6B post (n=142,135,142,140) | 134 | 127 | 135 | 138
  Opsono-7F pre (n=111,122,115,104) | 109 | 117 | 109 | 42
  Opsono-7F post (n=140,137,139,112) | 140 | 137 | 139 | 53
  Opsono-9V pre (n=133,133,130,130) | 131 | 130 | 122 | 126
  Opsono-9V post (n=143,139,143,137) | 143 | 139 | 143 | 137
  Opsono-14 pre (n=121,125,114,125) | 115 | 116 | 107 | 124
  Opsono-14 post (n=137,138,138,134) | 137 | 138 | 138 | 134
  Opsono-18C pre (n=126,118,123,123) | 45 | 54 | 34 | 35
  Opsono-18C post (n=121,129,121,114) | 121 | 127 | 121 | 110
  Opsono-19F pre (n=127,135,134,134) | 102 | 110 | 95 | 29
  Opsono-19F post (n=137,137,139,133) | 133 | 132 | 139 | 131
  Opsono-23F pre (n=132,136,128,137) | 121 | 120 | 105 | 124
  Opsono-23F post (n=145,143,146,143) | 145 | 143 | 146 | 143

9. Secondary Outcome: Number of Subjects With Cross-reactive Pneumococcal Serotype Antibody Concentrations Above the Cut-off Value
Description: Anti-pneumococcal antibody cut-off value assessed was 0.05 microgram per milliliter (µg/mL).
  The cross-reactive pneumococcal serotypes assessed include 6A and 19A.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 157 | 153 | 160 | 152
subjects
  Anti-6A pre (n=145,144,144,149) | 126 | 120 | 119 | 110
  Anti-6A post (n=156,152,159,152) | 152 | 145 | 149 | 148
  Anti-19A pre (n=145,153,145,151) | 130 | 138 | 121 | 87
  Anti-19A post (n=157,153,160,152) | 154 | 151 | 155 | 149

10. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes Above the Cut-off Value
Description: Anti-pneumococcal antibody cut-off value assessed was ≥ 8.
  The cross-reactive pneumococcal serotypes assessed include 6A and 19A.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 133 | 138 | 136 | 134
subjects
  Opsono-6A pre (n=108,110,106,110) | 68 | 66 | 73 | 62
  Opsono-6A post (n=127,128,128,122) | 116 | 119 | 117 | 119
  Opsono-19A pre (n=133,138,136,134) | 4 | 11 | 4 | 2
  Opsono-19A post (n=124,132,130,123) | 77 | 75 | 50 | 29

11. Secondary Outcome: Number of Subjects With Anti-protein D Antibody Concentrations Above the Cut-off Value
Description: Anti-protein D antibody cut-off value assessed was ≥ 100 Enzyme-Linked Immuno Sorbent Assay (ELISA) unit per milliliter (EL.U/mL).
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 158 | 153 | 160 | 148
subjects
  Pre (n=147,153,147,146) | 144 | 147 | 138 | 59
  Post (n=158,152,160,148) | 158 | 151 | 160 | 66

12. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Titer Above the Cut-off Value
Description: Meningococcal serogroup C serum bactericidal assay titer cut-off value assessed was ≥ 8.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 89 | 84 | 79 | 78
subjects
  Pre (n=68,65,66,78) | 57 | 62 | 62 | 68
  Post (n=89,84,79,76) | 89 | 84 | 79 | 76

13. Secondary Outcome: Number of Subjects With Anti-meningococcal Polysaccharide C Antibody Concentrations Above the Cut-off Value
Description: Anti-meningococcal polysaccharide C antibody cut-off value assessed was ≥ 0.3 µg/mL.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 156 | 149 | 159 | 149
subjects
  Pre (n=126,124,125,135) | 95 | 82 | 105 | 102
  Post (n=156,149,159,149) | 156 | 149 | 159 | 149

14. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate Antibody Concentrations Above the Cut-off Value
Description: Anti-polyribosyl-ribitol phosphate antibody cut-off value assessed was ≥ 0.15 µg/mL.
Time Frame: Before (pre) and one month after (post) the booster administration
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Number analyzed (Participants) | 157 | 153 | 160 | 152
subjects
  Pre (n=147,144,150,148) | 122 | 128 | 145 | 143
  Post (n=157,153,160,152) | 157 | 153 | 160 | 152

ADVERSE EVENTS:
Arm/Group | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Serious Adverse Events (participants affected / at risk) | 15 | 9 | 13 | 13
Other Adverse Events (participants affected / at risk) | 297/359 | 303/363 | 302/358 | 287/357
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ | Prevenar™ + Menitorix™
Gastroenteritis (Infections and infestations) | 2/359 | 4/363 | 2/358 | 3/357
Pneumonia (Infections and infestations) | 2/359 | 1/363 | 0/358 | 3/357
Febrile convulsion (Nervous system disorders) | 0/359 | 1/363 | 2/358 | 2/357
Gastroenteritis rotavirus (Gastrointestinal disorders) | 4/359 | 0/363 | 1/358 | 0/357
Bronchopneumonia (Infections and infestations) | 1/359 | 1/363 | 0/358 | 2/357
Bronchitis (Infections and infestations) | 1/359 | 0/363 | 1/358 | 1/357
Pharyngitis (Infections and infestations) | 0/359 | 1/363 | 2/358 | 0/357
Thermal burn (Injury, poisoning and procedural complications) | 2/359 | 0/363 | 1/358 | 0/357
Diarrhoea (Gastrointestinal disorders) | 0/359 | 0/363 | 0/358 | 2/357
Gastritis (Gastrointestinal disorders) | 1/359 | 1/363 | 0/358 | 0/357
Acute tonsillitis (Infections and infestations) | 0/359 | 0/363 | 1/358 | 0/357
Arthritis (Musculoskeletal and connective tissue disorders) | 0/359 | 0/363 | 1/358 | 0/357
Bronchpneumopathy (Respiratory, thoracic and mediastinal disorders) | 0/359 | 0/363 | 1/358 | 0/357
Breath holding (Psychiatric disorders) | 0/359 | 0/363 | 1/358 | 0/357
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0/359 | 0/363 | 1/358 | 0/357
Concussion (Injury, poisoning and procedural complications) | 0/359 | 0/363 | 0/358 | 1/357
Dehydration (Metabolism and nutrition disorders) | 1/359 | 0/363 | 0/358 | 0/357
Electric shock (Injury, poisoning and procedural complications) | 1/359 | 0/363 | 0/358 | 0/357
Epilepsy (Nervous system disorders) | 0/359 | 0/363 | 1/358 | 0/357
Laryngitis (Infections and infestations) | 0/359 | 0/363 | 0/358 | 1/357
Pyelonephritis acute (Infections and infestations) | 0/359 | 0/363 | 0/358 | 1/357
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/359 | 0/363 | 1/358 | 0/357
Salmonellosis (Infections and infestations) | 1/359 | 0/363 | 0/358 | 0/357
Tracheitis (Infections and infestations) | 1/359 | 0/363 | 0/358 | 0/357
Upper respiratory tract infection (Infections and infestations) | 0/359 | 1/363 | 0/358 | 0/357
Viral infection (Infections and infestations) | 0/359 | 1/363 | 0/358 | 0/357
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/359 | 1/363 | 0/358 | 0/357
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK's 10-valent Pneumococcal Vaccine 1024850A + Meningitec™ (N=359) | GSK's 10-valent Pneumococcal Vaccine 1024850A + NeisVac-C™ (N=363) | GSK's 10-valent Pneumococcal Vaccine 1024850A + Menitorix™ (N=358) | Prevenar™ + Menitorix™ (N=357)
Upper respiratory tract infection (Infections and infestations) | 6 | 19 | 14 | 18
Pain (General disorders) | 196 | 195 | 193 | 165
Redness (General disorders) | 194 | 183 | 186 | 173
Swelling (General disorders) | 162 | 148 | 150 | 134
Drowsiness (General disorders) | 124 | 142 | 139 | 105
Fever (General disorders) | 109 | 122 | 105 | 108
Irritability (General disorders) | 170 | 190 | 191 | 157
Loss of appetite (General disorders) | 101 | 99 | 112 | 93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.